CLINICAL TRIAL: NCT04655053
Title: Intervention for Self-regulation of Goals Related to Physical Exercise in People With Fibromyalgia: Motivational and Volitional Components
Brief Title: Intervention for Self-regulation to Physical Exercise in People With Fibromyalgia
Acronym: IAMEFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, María de los Ángeles Pastor Mira, Professor. Principal Investigator, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PSI2016-79566-C2-1-R
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; walking exercise; implementation intentions; self-regulation; pain catastrophizing; women
MeSH Terms: conditions — Fibromyalgia; Self-Control | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Intervention Model Description: Self-regulation condition (between-factor): Goal intention condition (IC), implementation intention condition focused on behavior initiation (IIC-Behavior), implementation intention condition focused on goal preference management (IIC-Motivational).
  Pain catastrophizing (within factor): Low (equal or less 31 score on this variable) and high (more than 31 score in this variable)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Goal intention condition (Active Comparator): Participants in this condition are asked to form the goal condition: "I will walk as fast as I can for as long as I can"
  Interventions: Behavioral: Goal intention
- Implementation intention (behavior initiation) condition (Experimental): Participants in this condition are asked to form the same goal intention ( "I will walk as fast as I can for as long as I can") and add the if-then plan ("and if I do the task, then I will walk as much as I can!")
  Interventions: Behavioral: Implementation intention to initiate the behavior
- Implementation intention (goal preference management) condition (Experimental): Participants in this condition are asked to form the same goal intention ( "I will walk as fast as I can for as long as I can") and add the if-then plan ("and if at this moment I prefer not to walk because of my pain (or fatigue; depending on person), then I will accept that I have this difficulty and I will walk as much as I can!)
  Interventions: Behavioral: Implementation intention to manage the goal preference (avoiding behavior or not)

INTERVENTIONS:
Behavioral: Goal intention — Researcher instructs participants to adopt and learn the goal intention requesting them to write it three times and verbally repeat once.
  Arms: Goal intention condition
Behavioral: Implementation intention to initiate the behavior — Researcher instructs participants to adopt and learn the goal intention and the plan requesting them to write it three times and verbally repeat once.
  Arms: Implementation intention (behavior initiation) condition
Behavioral: Implementation intention to manage the goal preference (avoiding behavior or not) — Researcher instructs participants to adopt and learn the goal intention and the plan requesting them to write it three times and verbally repeat once.
  Arms: Implementation intention (goal preference management) condition

SUMMARY:
This work is part of a broader research with women with fibromyalgia. The aim of this study is to establish the effectiveness of implementation intentions to manage the preference for avoiding pain and fatigue and stop walking exercise, versus to maintain the approximate behavior (walking), taking into account high and low pain catastrophizing conditions.

DETAILED DESCRIPTION:
Fibromyalgia is a widespread and diffuse musculoskeletal chronic pain problem not associated with inflammatory or degenerative changes, often accompanied by fatigue and sleep problems, in addition to anxiety, depression and cognitive dysfunction. Its prevalence in Europe for adults is estimated at 2.5% with a higher proportion of women. The treatment incorporates physical activity and exercise as one of its therapeutic aims has shown positive effects on health outcomes.However, it has been reported that women with fibromyalgia are less active than others with similar socio-demographic characteristics.Theories of behavioral self-regulation that taking into account motivational and volitional processes (implementation intentions) provide a conceptual framework to work with the incorporation and maintenance of the exercise, helping these people to create strong goals and handle the different self-regulation problems that can arise. These include the ones related to the preference for avoidance goals (pain or fatigue avoidance) against performing or keep doing an activity (walking exercise). This work searches to help women with fibromyalgia to manage the above mentioned inhibitors to incorporate and maintain long-term physical exercise walking. We consider the heterogeneity of people with fibromyalgia in pain catastrophizing, which makes necessary to adapt interventions aimed to promote physical exercise.

We expect participants with high catastrophizing and implementation intentions to control the preference for avoiding pain or fatigue will walk more time than the other conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women with fibromyalgia attended the Fibromyalgia Unit of the Valencian Community (Hospital of San Vicente del Raspeig, Alicante)
* Within the age limits

Exclusion Criteria:

* Comorbidity that prevents walking
* Those related to the 6MWT application protocol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Time of walking | Immediately after the experimental intervention
  The six-minutes walk test (6MWT) test is adapted to simulate a behavioural maintenance scenario of the walking exercise. Thus, the measure is the time of walking (maximum of 30m)

SECONDARY OUTCOMES:
Perceived exertion | Immediately after the experimental intervention
  Score on the Borg Rating of Perceived Exertion Scale anchored at 10 (Borg: 0=Not exertion at all; 10=Maximal). Higher scores mean higher perceived exertion.
Physical activity intensity | Immediately after the experimental intervention
  Percentage of participants with moderate physical activity according to the accelerometer.
Walking speed | Immediately after the experimental intervention
  Speed mean in each experimental group

CONTACTS AND LOCATIONS:
Overall Officials: María-Ángeles Pastor-Mira, PhD, Principal Investigator — Universidad Miguel Hernández
Locations (1):
- Hospital de San Vicente del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No